CLINICAL TRIAL: NCT01536431
Title: Phase 1b Study of Proinsulin (PI) Peptide Immunotherapy in New-Onset Type 1 Diabetes
Brief Title: Safety Study to Assess Whether Proinsulin Peptide Injections Can Slow or Stop the Body Damaging Its Own Insulin-making Cells in the Pancreas in Patients Newly Diagnosed With Type 1 Diabetes
Acronym: MonoPepT1De
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Diabetes Vaccine Development Centre (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Professor Colin Dayan, Professor, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPON817-10; 2007-003759-35 (EudraCT Number); 66760879 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-02-14; First posted 2012-02-22 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pro insulin peptide (Experimental): Patients will receive 10 micro gr of the peptide every 2 weeks (12 doses).
  Interventions: Drug: Pro insulin peptide
- Pro insulin peptide & saline (Active Comparator): Patients will receive 10 micro gr of the peptide monthly (ever 4 weeks, 6 doses) and saline injections monthly alternating with the peptide (2 weeks interval between the drug and saline).
  Interventions: Drug: Pro insulin peptide
- Saline (Placebo Comparator): Patients will receive 0 micro gr of peptide, but have saline injections every 2 weeks (controls)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Pro insulin peptide — Patients will receive 10 micro gr of the peptide every 2 weeks (12 doses).
  Arms: Pro insulin peptide
Drug: Pro insulin peptide — Patients will receive 10 micro gr of the peptide monthly (ever 4 weeks, 6 doses) and saline injections monthly alternating with the peptide (2 weeks interval between the drug and saline).
  Arms: Pro insulin peptide & saline
Drug: Saline — Patients will receive 0 micro gr of peptide, but have saline injections every 2 weeks (controls).
  Arms: Saline

SUMMARY:
The purpose of this study is to address the safety issue of whether, in patients with newly-diagnosed diabetes who still make some insulin, proinsulin peptide therapy adversely affects the rate of damage to the insulin making cells.

DETAILED DESCRIPTION:
Type 1 Diabetes (also known as insulin-dependent diabetes) is caused by destruction of the insulin producing cells (Beta Cells) in the pancreas. Our group is interested in how this destruction could be stopped or reversed, as this may lead to development of a new generation of diabetes treatments which can prevent or slow down the damage, reducing or possibly even removing there need for insulin injections.

In a previous study we examined the safety of our novel approach to this problem, proinsulin (PI) peptide immunotherapy, in longstanding diabetes patients (diagnosed more than 5 years before), and found it to be well tolerated and free of major hypersensitivity reactions. However, it remains theoretically possible that this form of immunotherapy could make the immune reaction to the insulin making cells worse rather than better.

This cannot be studied directly in longstanding patients as they have no or almost no insulin making cells left.

So,the principle objective of the current study is to address the safety issue of whether, in patients with newly-diagnosed diabetes who still make some insulin, proinsulin peptide therapy adversely affects the rate of damage to the insulin making cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years.
2. If female, must be (as documented in patient notes):

   * postmenopausal (at least 1 year without spontaneous menses)
   * surgically sterile (tubal ligation or hysterectomy at least 6 months prior to enrolment)
   * using acceptable contraception (e.g., oral, intramuscular, or implanted hormonal contraception) at least 3 months prior to enrolment
   * have a sexual partner with non-reversed vasectomy (with confirmed azoospermia)
   * be using 1 barrier method with the use of a spermicide(e.g., condom, diaphragm or cap)
   * have placement of a intra-uterine device
3. If male, must be:

   * using a barrier method of contraception (condom) with the use of a spermicide
   * have a sexual partner using one of the methods in point 2 above or
   * have a non-reversed vasectomy (with confirmed azoospermia),
4. Diagnosis of Type 1 diabetes within the last 100 days (dated from the first insulin injection).
5. Possession of *0401 allele at the HLA-DRB1 gene locus
6. At least one positive islet cell autoantibody (ie anti-GAD65, antibodies to insulinoma-associated antigen-2 (IA-2) or zinc transporter 8 (ZnT8)).
7. Peak insulin C-peptide >200 pmol/L (at any time point after stimulation with Mixed Meal Tolerance Test).
8. Written and witnessed informed consent to participate.

Exclusion Criteria:

1. Females who are pregnant, breast-feeding or not using adequate forms of contraception.
2. Use of immunosuppressive or immunomodulatory therapies, including systemic steroids within 1 month prior to randomisation and any monoclonal antibody therapy given for any indication.
3. Any other medical condition which, in the opinion of investigators, could affect the safety of the subject's participation.
4. Recent subject's involvement in other research studies which, in the opinion of investigators, may adversely affect the safety of the subjects or the results of the study.
5. Subjects should not have had immunisations with live or killed vaccines or allergic desensitisation procedures less than 1 month prior to their first treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety | 3 years
  To address the safety issue of whether, in patients with newly-diagnosed diabetes who still make some insulin, proinsulin peptide therapy adversely affects the rate of damage to the insulin making cells.

SECONDARY OUTCOMES:
Allergy and hypersensitivity | 3 years
  To confirm that PI peptide treatment does not induce allergy or hypersensitivity and has a good safety profile in new-onset type 1 diabetes patients.
Safety of frequent dosing | 3 years
  To explore the safety of extending peptide treatment to more frequent dosing (2-weekly) and for a longer time period (6 months)
Protective effects of insulin preservation | 3 years
  To provide preliminary data on any protective effect on preservation of insulin production after 1 year of treatment
T cell (immune) response to islet cell antigens | 3 years
  To provide preliminary data on changes in the T cell (immune) response to islet cell antigens in newly-diagnosed patients following PI peptide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Peakman, MBBS BSc MSc PhD FRCP, Study Director — King's College Hospital NHS Trust
Locations (5):
- United Kingdom (5):
  - Countess of Chester, Chester, England
  - Bristol Royal Infirmary, Bristol
  - University Hospital of Wales, Cardiff
  - Guy's Hospital, London
  - Royal Victoria Hospital, Newcastle